CLINICAL TRIAL: NCT03286426
Title: Ocular Screening in Children and Young Adults at Risk for Increased Intracranial Pressure
Acronym: ICP
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: COVID
Sponsor: Duke University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: Pro00083580
Record Dates: First submitted 2017-09-14; First posted 2017-09-18 (Actual); Results first posted 2022-02-15 (Actual); Last update posted 2022-02-15 (Actual); Status verified 2022-01

CONDITIONS: Intracranial Pressure Increase
Keywords: vision screening; portable fundus camera; acne medication
MeSH Terms: conditions — Intracranial Hypertension

STUDY DESIGN:
Intervention Model Description: All patients will have images taken of the back of the eye with a portable fundus camera. If able, visual acuity and color vision will be checked.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Vision/Eye Screening (Experimental): Image of back of each eye along with color vision and visual acuity assessment if able.
  Interventions: Diagnostic Test: Pictor

INTERVENTIONS:
Diagnostic Test: Pictor — The back of each eye will be imaged with Pictor. Visual acuity and color vision will be checked if patient able to cooperate with exam.
  Other Names: portable fundus camera

SUMMARY:
The purpose of this study is to evaluate the vision and posterior segment of eyes in children and young adults less than 22 years of age with risk, suspicion, or past medical history significant for elevated intracranial pressure (ICP). Patients will have visual acuity and color vision tested. Assessment of the posterior segment will involve using a non-invasive (non-contact) imaging technique (i.e. a portable fundus camera in clinic and hospital settings).

DETAILED DESCRIPTION:
The need for non-invasive evaluation of ICP is an active area of study. The current gold standard is intraventricular or intraparenchymal catheters but these are invasive, expensive, and require sedation; and thus the need for an effective non-invasive screening tool. The utility of funduscopy in identifying processes affecting ICP has long been recognized, i.e. papilledema, ocular venous engorgement, blurring of the optic disk. Studies have demonstrated that funduscopy may have a role in the qualitative assessment of increased ICP as a highly sensitive test. However, conventional bedside funduscopy does not allow for image capture and may necessitate pupillary dilation. Portable fundus cameras address these issues, allowing image capture and storage and the potential for non-mydriatic imaging, i.e. imaging without dilation of eyes. And as demonstrated in a recent study, portable fundus cameras are efficient (median exam time was 3 minutes and 24 seconds in a pediatric Emergency Department).

Additionally, ICP screening in asymptomatic patients remains limited. Patients being treated with medications for acne, specifically tetracyclines (e.g. minocycline and doxycycline), retinol, and isotretinol, are at particular risk for increased ICP but often are not identified until they are symptomatic (i.e. headaches, visual loss, papilledema). Symptom onset has been documented from 2 weeks up to 1 year from drug initiation. The percentage of patients with subclinical asymptomatic disease is unclear. This study would allow us to describe the presence of subclinical disease in our population and the role/utility of routine non-invasive screening methods.

ELIGIBILITY:
Inclusion Criteria:

* Capable and willing to provide consent
* Less than 22 years of age
* History of or suspicion for elevated ICP or starting/currently taking high-risk medications associated with increased risk for elevated ICP

Exclusion Criteria:

* Unable or unwilling to give consent
* Over 21 years of age

Max Age: 21 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 3 (Actual)
Dates: Start 2017-10-26 (Actual); Primary Completion 2018-12-08 (Actual); Study Completion 2018-12-08 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sarah K Jones, Study Director — Duke University
Locations (1):
- Duke UMC, Durham, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Xu W, Gerety P, Aleman T, Swanson J, Taylor J. Noninvasive methods of detecting increased intracranial pressure. Childs Nerv Syst. 2016 Aug;32(8):1371-86. doi: 10.1007/s00381-016-3143-x. Epub 2016 Jun 28. PMID 27351182
- [Background] Roberts E, Morgan R, King D, Clerkin L. Funduscopy: a forgotten art? Postgrad Med J. 1999 May;75(883):282-4. doi: 10.1136/pgmj.75.883.282. PMID 10533632
- [Background] Sit M, Levin AV. Direct ophthalmoscopy in pediatric emergency care. Pediatr Emerg Care. 2001 Jun;17(3):199-204; quiz 205-7. doi: 10.1097/00006565-200106000-00013. PMID 11437148
- [Background] Petrushkin H, Barsam A, Mavrakakis M, Parfitt A, Jaye P. Optic disc assessment in the emergency department: a comparative study between the PanOptic and direct ophthalmoscopes. Emerg Med J. 2012 Dec;29(12):1007-8. doi: 10.1136/emermed-2011-200038. Epub 2011 Oct 13. PMID 21998469
- [Background] Golshani K, Ebrahim Zadeh M, Farajzadegan Z, Khorvash F. Diagnostic Accuracy of Optic Nerve Ultrasonography and Ophthalmoscopy in Prediction of Elevated Intracranial Pressure. Emerg (Tehran). 2015 Spring;3(2):54-8. PMID 26495382
- [Background] Day LM, Wang SX, Huang CJ. Nonmydriatic Fundoscopic Imaging Using the Pan Optic iExaminer System in the Pediatric Emergency Department. Acad Emerg Med. 2017 May;24(5):587-594. doi: 10.1111/acem.13128. Epub 2017 Mar 24. PMID 27801997
- [Background] Friedman DI. Medication-induced intracranial hypertension in dermatology. Am J Clin Dermatol. 2005;6(1):29-37. doi: 10.2165/00128071-200506010-00004. PMID 15675888
- [Background] Chiu AM, Chuenkongkaew WL, Cornblath WT, Trobe JD, Digre KB, Dotan SA, Musson KH, Eggenberger ER. Minocycline treatment and pseudotumor cerebri syndrome. Am J Ophthalmol. 1998 Jul;126(1):116-21. doi: 10.1016/s0002-9394(98)00063-4. PMID 9683157

RESULTS

PARTICIPANT FLOW:
Groups:
- Vision/Eye Screening: Image of back of each eye along with color vision and visual acuity assessment if able.
  Vision/Eye screening: The back of each eye will be imaged with Pictor. Visual acuity and color vision will be checked if patient able to cooperate with exam.
Period: Overall Study
Arm/Group | Vision/Eye Screening
Started | 3
Completed | 0
Not Completed | 3
Not completed — Physician Decision | 3

BASELINE CHARACTERISTICS:
Arm/Group | Vision/Eye Screening
Number analyzed (Participants) | 3
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3
  Between 18 and 65 years | 0
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: months] | 59 (75)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 2
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0
  Not Hispanic or Latino | 3
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 1
  White | 2
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 3

OUTCOME MEASURES:

1. Primary Outcome: Changes in Posterior Segment as Measured by Fundus Camera
Time Frame: Each visit (up to 1 hour/visit) every 3 months for 1 year from signed consent
Population: Data not collected as only one visit occurred and a change could not be measured.
Arm/Group | Vision/Eye Screening
Number analyzed (Participants) | 0

2. Primary Outcome: Changes in Visual Acuity
Time Frame: Each visit (up to 1 hour/visit) every 3 months for 1 year from signed consent
Population: Data not collected as only one visit occurred and a change could not be measured.
Arm/Group | Vision/Eye Screening
Number analyzed (Participants) | 0

3. Primary Outcome: Changes in Color Vision as Measured by Standard Clinical Exam (i.e. Ishihara Testing)
Time Frame: Each visit (up to 1 hour/visit) every 3 months for 1 year from signed consent
Population: Data not collected as only one visit occurred and a change could not be measured.
Arm/Group | Vision/Eye Screening
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: At baseline visit as only one visit occurred for each subject.
Description: All-Cause Mortality, Serious, and Other (Not Including Serious) Adverse Events were not monitored/assessed as there was only one visit per subject for this study.
Arm/Group | Vision/Eye Screening
All-Cause Mortality (participants affected / at risk) | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-11-14): https://cdn.clinicaltrials.gov/large-docs/26/NCT03286426/Prot_SAP_000.pdf